CLINICAL TRIAL: NCT05148910
Title: Satisfaction, Continuity, and Bleeding Patterns in Patients With Breast Cancer Using Copper and Silver Intrauterine Device (IUD) Compared to Copper IUD: a Randomized Clinical Trial
Brief Title: Breast Cancer and Intrauterine Contraception
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Edson Santos Ferreira-Filho (Unknown); Nilson Roberto de Melo (Unknown); Isabel Cristina Esposito Sorpreso (Unknown); José Maria Soares Júnior (Unknown); José Roberto Filassi (Unknown); Kátia Cândido Carvalho (Unknown); Walter da Silva Pinheiro (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26272819.3.0000.0068
Record Dates: First submitted 2021-09-03; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Contraception
Keywords: breast cancer; contraception; intrauterine device
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copper IUD (TCu380A) (Active Comparator): Women receiving an intrauterine device (IUD) containing 380mm² of copper.
  Interventions: Device: Copper IUD (TCu380A)
- Silver and copper IUD (TCu380Ag) (Experimental): Women receiving an intrauterine device (IUD) containing 380mm² of copper with a silver core.
  Interventions: Device: Silver and copper IUD (TCu380Ag)

INTERVENTIONS:
Device: Silver and copper IUD (TCu380Ag) — An intrauterine device containing 380mm² of copper with a silver core.
  Arms: Silver and copper IUD (TCu380Ag)
Device: Copper IUD (TCu380A) — An intrauterine device containing 380mm² of copper.
  Arms: Copper IUD (TCu380A)

SUMMARY:
The present work seeks an alternative to the copper IUD for contraception in breast cancer patients, evaluating the satisfaction and continuity of the copper and silver IUD, as well as the quality of life, compared to the copper IUD, especially in the regarding the menstrual bleeding pattern of these patients and possible mechanisms that justify such differences. A randomized (1:1) controlled clinical trial is proposed. Women between 18 and 45 years of age, diagnosed with breast carcinoma through histopathological study, who have had at least one vaginal sexual intercourse in life and wish to use intrauterine contraception will be included.

DETAILED DESCRIPTION:
A randomized (1:1) controlled clinical trial is proposed. Women aged 18 to 45 years, diagnosed with breast carcinoma through histopathological study will be included. The study will be conducted at the Family Planning Outpatient Clinic of the Division of Gynecology, Hospital das Clínicas, Faculty of Medicine, University of São Paulo (HC-FMUSP). The primary source of recruitment of patients will be the Mastology Outpatient Clinic of the São Paulo Cancer Institute "Octavio Frias de Oliveira" (ICESP). After selecting the patients and signing the informed consent form (ICF), research participants will receive specific reproductive counseling, with guidance on all contraceptive methods available and appropriate for their health condition.

To minimize selection bias, subjects will be randomized to one of two groups: 1) Copper IUD (TCu380A); or 2) Copper and silver IUD (TCu380Ag), in a proportion 1:1. The randomization sequence was generated using the website http://www.randomization.com. Information on which treatment each woman will be assigned will be kept in a sealed, opaque envelope identified with a number. The envelope will only be opened after the participant has signed the ICF. Once the allocation is made, it cannot be changed. Only the professional who inserts the device knows the type of IUD. Patients will not know which type of IUD they will use to minimize performance bias, i.e., they will be blinded to the nature of the inserted device. Blinding will not be revealed until the end of the study.

Patients will be evaluated 3, 6 and 12 months after IUD insertion. This follow-up will be carried out at the Family Planning Clinic of the Gynecology Division at HC-FMUSP. After informed consent, patients will be asked about their current age, occupation, scholarship, ethnicity/race, date of cancer diagnosis, age at menarche and first sexual intercourse, number of lifetime partners, sexual orientation, number of pregnancies, deliveries and abortions, duration of breastfeeding, age of first and last birth, date of last menstruation, lifetime use of hormonal and emergency contraception, condom use, pregnancy desire after cancer treatment, comorbidities, type of surgery (conservative or mastectomy), current use of SERMS (selective estrogen receptor modulators; tamoxifen or raloxifene), aromatase inhibitors and anticoagulants, smoking (quantity and duration), alcoholism (frequency and dose), physical activity (type, time and duration), family history of malignant neoplasms. Tumor staging (TNM) and the immunohistochemical panel will also be recorded. In addition, the menstrual bleeding pattern will be questioned (through the recall of the last three months), including the interval between cycles, number of days of menstruation and number of pads or tampons used and the occurrence of menstrual cramps and the use of analgesics during the menstrual period. At inclusion, weight (kg), height (cm), blood pressure (mmHg), waist circumference (cm) and hip (cm) will be measured. At the time of the gynecological examination, Pap smear and endocervical swab for Chlamydia trachomatis (PCR) will be collected. Blood samples will be collected for the following laboratory tests: blood count and serum levels of FSH, estradiol, iron, ferritin, transferrin, and total iron binding capacity. Dependent variables will be considered: continuation rates, satisfaction, quality of life, pregnancy, rates, and reasons for discontinuation, with an emphasis on abnormal uterine bleeding. The independent variable will be the IUD type. The control variables will be the aforementioned clinical and sociodemographic parameters.

After being included in the study, the IUD will be inserted by a trained professional, if there is assurance that the patient is not pregnant. Hysterometry (in centimeters) will be measured and recorded before insertion of the IUD. After insertion, the pain attributed to the procedure will be questioned, in a global way, through a visual analogue pain scale. For greater uniformity, all IUDs will be inserted on an outpatient basis, without local anesthesia and/or sedation.

After 30 to 90 days of insertion, patients will undergo a physical examination (visualization of the IUD thread) and transvaginal ultrasound to verify if the IUD is in situ.

Patients will be evaluated 3, 6 and 12 months after IUD insertion. The clinical performance of the IUDs will be evaluated, including pregnancy, infection, perforation, expulsion, continuity of use, reasons for discontinuation, satisfaction with the method, menstrual bleeding pattern (PABC) and laboratory tests (blood count and serum levels of FSH, estradiol, iron, ferritin, transferrin, and total iron binding capacity). The PABC (pictorial blood loss assessment chart) tool will be used to collect information about menstrual bleeding. Increased uterine bleeding will be defined as a PABC score greater than 100 and/or bleeding duration greater than 7 days and/or by the woman's subjective perception of increased menstrual flow.

To assess quality of life, the Medical Outcomes Study 36-Item Short-Form Healty Survey (SF-36) questionnaire will be used. The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) will also be included.

The collected data will be systematized in confidential spreadsheets for statistical analysis supervised by a qualified statistician. Quantitative description of the data (mean, median, standard deviation and relative frequency) will be performed and the analyzes will be performed using appropriate tests for each type of variable: quantitative variables will be analyzed by t test (parametric) or Mann-Whitney (non-parametric), according to the normality of the distribution; and categorical variables will be analyzed by chi-square (χ²) or Fisher's exact test, according to the number of observed events. The normality of data distribution will be evaluated using the Kolmogorov-Smirnov and Shapiro-Wilk tests. The time for the occurrence of events will be described in Kaplan-Meier curves and possible differences will be analyzed using the log-rank test and using proportional hazards models (Cox regression) using clinical-demographic and laboratory variables. The results will be reported as Relative Risk (RR), Odds Ratio (OR) and Hazard Ratios (HR), with 95% confidence intervals (95%CI). Both intention-to-treat and per-protocol analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast carcinoma through histopathological study
* At least one vaginal sexual intercourse in life
* Wish to use intrauterine contraception

Exclusion Criteria:

* Currently pregnant women
* Postmenopausal women
* Hysterectomized and/or bilaterally ovariectomized women
* Abortion less than four weeks
* Childbirth less than six weeks
* Known endometrial cavity changes
* Severe anemia (hemoglobin < 8 g/dL)
* Severe thrombocytopenia
* Acute purulent cervicitis
* Current endometritis
* Acute pelvic inflammatory disease
* Genital tuberculosis
* Genital bleeding of unknown cause
* Cervical or endometrial cancer
* Wilson's disease
* Cognitive or psychiatric disorder that makes adherence to the study protocol unfeasible
* Tubal ligation
* Women who do not agree to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Continuity | 3 months
  Number of women that decide to continue using the method assigned
Continuity | 6 months
  Number of women that decide to continue using the method assigned
Continuity | 12 months
  Number of women that decide to continue using the method assigned
Subjects' Satisfaction | 3 months
  Number of women who are satisfied with the method assigned
Subjects' Satisfaction | 6 months
  Number of women who are satisfied with the method assigned
Subjects' Satisfaction | 12 months
  A likert Scale including the question "Are you satisfied with the IUD?" and the answers: extremely satisfied; very satisfied; a little satisfied; neither satisfied nor dissatisfied; a little dissatisfied; very dissatisfied; extremely dissatisfied
Bleeding pattern | 3 months
  Number of days of bleeding, punctuation through pictorial assessment blood chart
Bleeding pattern | 6 months
  Number of days of bleeding, punctuation through pictorial assessment blood chart
Bleeding pattern | 12 months
  Number of days of bleeding, punctuation through pictorial assessment blood chart

SECONDARY OUTCOMES:
Quality of life (SF-36) | 12 months
  Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
Quality of life (EORTC QLQ-C30) | 12 months
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Complete blood count | Baseline
  Complete blood count
Complete blood count | 6 months
  Complete blood count
Complete blood count | 12 months
  Complete blood count
Serum iron | Baseline
  Serum iron
Serum iron | 6 months
  Serum iron
Serum iron | 12 months
  Serum iron
Ferritin level | Baseline
  Ferritin level
Ferritin level | 6 months
  Ferritin level
Ferritin level | 12 months
  Ferritin level
Transferrin level | Baseline
  Transferrin level
Transferrin level | 6 months
  Transferrin level
Transferrin level | 12 months
  Transferrin level
Total iron binding capacity | Baseline
  Total iron binding capacity
Total iron binding capacity | 6 months
  Total iron binding capacity
Total iron binding capacity | 12 months
  Total iron binding capacity

CONTACTS AND LOCATIONS:
Overall Officials: Edmund C Baracat, PhD, Principal Investigator — Faculdade de Medicina FMUSP, Universidade de Sao Paulo, Sao Paulo, Brazil.
Locations (1):
- Hospital das Clínicas HCFMUSP, Faculdade de Medicina, Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) might be available to other researchers after publication of all planned results by research team.